CLINICAL TRIAL: NCT06635876
Title: Piloting an Online Emergency Preparedness Toolkit for Caregivers Preparing for Their Own Health Care Emergency
Brief Title: Caregivers Preparing for Their Own Health Care Emergency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2180909; 1R21AG089840-01 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Caregiver Burden
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPT-C (Active Comparator): The EPT-C group will receive two coaching sessions to assist with the completion of the EPT.
  Interventions: Behavioral: Coaching Sessions
- EPT-A (No Intervention): The EPT-A group will be responsible for completing the EPT alone, without coaching sessions.

INTERVENTIONS:
Behavioral: Coaching Sessions — The coach will use motivational interviewing techniques to:
  1. To assist and guide the caregiver to establish a standby caregiver relationship
  2. To assist and guide the caregiver as to how to use the EPT
  Arms: EPT-C

SUMMARY:
The proposed research will develop and test an online Emergency Preparedness Toolkit to help caregivers prepare for their own unexpected health events. Caregivers of persons with dementia often ignore their own health needs as their primary focus is the care of the person with dementia. This can lead to a caregiver delaying their own care and subsequently emergent health events. The Emergency Preparedness Toolkit provides guidance to the caregiver as to how to identify and transfer care to a standby caregiver. The goal is to provide a caregiver with the security and comfort that the person with dementia will be well cared for while they care for their own health needs.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older at the time of signing the informed consent
* Must self-identify as the spouse or partner of the PWD
* Must provide some caregiving to a PWD
* Must live in the same dwelling as the PWD

Exclusion Criteria:

* Diagnosis of dementia
* Unable to use or does not have access to a computer
* Complete deafness or blindness and/or unable to use a telephone
* Condition that prevents them from performing caregiving duties or providing physical/emotional support to the PWD
* Unable to follow directions
* Unable to read or write in English
* Participation in prior study involving the EPT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Completion of the EPT six weeks from the baseline visit | Six weeks
  This will be measured using de-identified data from the EPT system.

SECONDARY OUTCOMES:
Identification and engagement of a standby caregiver six weeks from the baseline visit | Six weeks
  This will be measured using de-identified data from the EPT system.
Change in caregiver preparedness from baseline to Month 3 | Three months
  This will be measured using the Caregiver Preparedness Scale (CPS). Responses are rated from 0 to 4. The higher the score, the more prepared the caregiver feels for caregiver; the lower the score, the less prepared the caregiver feels.
Change in caregiver confidence from baseline to Month 3 | Three months
  This will be measured using a Likert scale of caregiver confidence from "completely confident" to "not at all confident". Responses will be grouped into two categories: confident (completely confident, fairly confident, or somewhat confident) or not confident (slightly confident or not at all confident).
Change in caregiving self-efficacy from baseline to Month 3 | Three months
  This will be measured using the Revised Scale for Caregiver Self-Efficacy (RSCSE). Responses are rated from 0 to 100. The higher the score, the more self-efficacious the caregiver feels about caregiving; the lower the score, the less self-efficacious the caregiver feels.
Qualitative data and theme identification from participant experience surveys and EPT-C coaching session recordings | Three months
  This will be measured using a qualitative descriptive approach and theme identification, based on participant experience surveys and EPT-C coaching session recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Boxer, MD, MS, Principal Investigator — University of California, Davis
Locations (1):
- University of California - Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brodaty H, Donkin M. Family caregivers of people with dementia. Dialogues Clin Neurosci. 2009;11(2):217-28. doi: 10.31887/DCNS.2009.11.2/hbrodaty. PMID 19585957
- [Background] Ornstein KA, Wolff JL, Bollens-Lund E, Rahman OK, Kelley AS. Spousal Caregivers Are Caregiving Alone In The Last Years Of Life. Health Aff (Millwood). 2019 Jun;38(6):964-972. doi: 10.1377/hlthaff.2019.00087. PMID 31158025
- [Background] Rykkje L, Tranvåg O. Caring for one's wife with dementia-at home: older husbands' experiences with managing challenges of everyday life. Sage Open. 2019;9(1):215824401983445. doi:10.1177/2158244019834453
- [Background] Perkins M, Howard VJ, Wadley VG, Crowe M, Safford MM, Haley WE, Howard G, Roth DL. Caregiving strain and all-cause mortality: evidence from the REGARDS study. J Gerontol B Psychol Sci Soc Sci. 2013 Jul;68(4):504-12. doi: 10.1093/geronb/gbs084. Epub 2012 Oct 2. PMID 23033358
- [Background] Tarlow BJ, Wisniewski SR, Belle SH, Rubert M, Ory MG, Gallagher-Thompson D. Positive aspects of caregiving: Contributions of the REACH project to the development of new measures for Alzheimer's caregiving. Res Aging. 2004;26(4):429-453. doi:10.1177/0164027504264493
- [Background] Pinquart M, Sorensen S. Correlates of physical health of informal caregivers: a meta-analysis. J Gerontol B Psychol Sci Soc Sci. 2007 Mar;62(2):P126-37. doi: 10.1093/geronb/62.2.p126. PMID 17379673
- [Background] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Background] Boxer RS, Daddato AE, Jessen A, Portz JD, Shetterly S. Hospitalizations of Caregivers Increases Risk of Hospitalization for Patients Living with Dementia. J Gen Intern Med. 2023 Feb;38(2):502-507. doi: 10.1007/s11606-022-07902-w. Epub 2022 Nov 14. No abstract available. PMID 36376629
- [Background] Whitlatch CJ, Orsulic-Jeras S. Meeting the Informational, Educational, and Psychosocial Support Needs of Persons Living With Dementia and Their Family Caregivers. Gerontologist. 2018 Jan 18;58(suppl_1):S58-S73. doi: 10.1093/geront/gnx162. PMID 29361068
- [Background] Pearce J, Forsyth W, Boyd R, Jackson GA. Empowering people with dementia: Rutherglen and Cambuslang Values History Project. Dementia. 2012;11(5):695-698. doi:10.1177/1471301211431364
- [Background] Mittelman MS, Haley WE, Clay OJ, Roth DL. Improving caregiver well-being delays nursing home placement of patients with Alzheimer disease. Neurology. 2006 Nov 14;67(9):1592-9. doi: 10.1212/01.wnl.0000242727.81172.91. PMID 17101889
- [Background] Yaffe K, Fox P, Newcomer R, Sands L, Lindquist K, Dane K, Covinsky KE. Patient and caregiver characteristics and nursing home placement in patients with dementia. JAMA. 2002 Apr 24;287(16):2090-7. doi: 10.1001/jama.287.16.2090. PMID 11966383
- [Background] Young HM, Bell JF, Whitney RL, Ridberg RA, Reed SC, Vitaliano PP. Social Determinants of Health: Underreported Heterogeneity in Systematic Reviews of Caregiver Interventions. Gerontologist. 2020 Feb 14;60(Suppl 1):S14-S28. doi: 10.1093/geront/gnz148. PMID 32057083
- [Background] Wawrziczny E, Berna G, Ducharme F, Kergoat MJ, Pasquier F, Antoine P. Modeling the Distress of Spousal Caregivers of People with Dementia. J Alzheimers Dis. 2017;55(2):703-716. doi: 10.3233/JAD-160558. PMID 27716667
- [Background] Turner RL, Reese-Melancon C, Harrington EE, Andreo M. Caregiving During the COVID-19 Pandemic: Factors Associated With Feelings of Caregiver Preparedness. J Appl Gerontol. 2023 Oct;42(10):2089-2099. doi: 10.1177/07334648231182242. Epub 2023 Jul 3. PMID 37395127
- [Background] Kasper JD, Freedman VA, Spillman BC, Wolff JL. The Disproportionate Impact Of Dementia On Family And Unpaid Caregiving To Older Adults. Health Aff (Millwood). 2015 Oct;34(10):1642-9. doi: 10.1377/hlthaff.2015.0536. PMID 26438739
- [Background] Pristavec T. The Burden and Benefits of Caregiving: A Latent Class Analysis. Gerontologist. 2019 Nov 16;59(6):1078-1091. doi: 10.1093/geront/gny022. PMID 29659788
- [Background] Waligora KJ, Bahouth MN, Han HR. The Self-Care Needs and Behaviors of Dementia Informal Caregivers: A Systematic Review. Gerontologist. 2019 Sep 17;59(5):e565-e583. doi: 10.1093/geront/gny076. PMID 29931147
- [Background] Oliveira D, Zarit SH, Orrell M. Health-Promoting Self-Care in Family Caregivers of People With Dementia: The Views of Multiple Stakeholders. Gerontologist. 2019 Sep 17;59(5):e501-e511. doi: 10.1093/geront/gnz029. PMID 30953585
- [Background] Mitchell SL, Teno JM, Kiely DK, Shaffer ML, Jones RN, Prigerson HG, Volicer L, Givens JL, Hamel MB. The clinical course of advanced dementia. N Engl J Med. 2009 Oct 15;361(16):1529-38. doi: 10.1056/NEJMoa0902234. PMID 19828530
- [Background] Sorensen S, Duberstein P, Gill D, Pinquart M. Dementia care: mental health effects, intervention strategies, and clinical implications. Lancet Neurol. 2006 Nov;5(11):961-73. doi: 10.1016/S1474-4422(06)70599-3. PMID 17052663
- [Background] Wang XR, Liu SX, Robinson KM, Shawler C, Zhou L. The impact of dementia caregiving on self-care management of caregivers and facilitators: a qualitative study. Psychogeriatrics. 2019 Jan;19(1):23-31. doi: 10.1111/psyg.12354. Epub 2018 Aug 7. PMID 30088311
- [Background] Acton GJ. Health-promoting self-care in family caregivers. West J Nurs Res. 2002 Feb;24(1):73-86. doi: 10.1177/01939450222045716. PMID 11829276
- [Background] Daddato AE, Dollar B, Lum HD, Burke RE, Boxer RS. Identifying Patient Readmissions: Are Our Data Sources Misleading? J Am Med Dir Assoc. 2019 Aug;20(8):1042-1044. doi: 10.1016/j.jamda.2019.04.028. Epub 2019 Jun 18. PMID 31227472
- [Background] Amjad H, Mulcahy J, Kasper JD, Burgdorf J, Roth DL, Covinsky K, Wolff JL. Do Caregiving Factors Affect Hospitalization Risk Among Disabled Older Adults? J Am Geriatr Soc. 2021 Jan;69(1):129-139. doi: 10.1111/jgs.16817. Epub 2020 Sep 22. PMID 32964422
- [Background] Gallagher-Thompson D, Choryan Bilbrey A, Apesoa-Varano EC, Ghatak R, Kim KK, Cothran F. Conceptual Framework to Guide Intervention Research Across the Trajectory of Dementia Caregiving. Gerontologist. 2020 Feb 14;60(Suppl 1):S29-S40. doi: 10.1093/geront/gnz157. PMID 32057080
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People for Change, 2nd Edition. 2nd ed. The Guilford Press; 2002:428.
- [Background] Archbold PG, Stewart BJ, Greenlick MR, Harvath T. Mutuality and preparedness as predictors of caregiver role strain. Res Nurs Health. 1990 Dec;13(6):375-84. doi: 10.1002/nur.4770130605. PMID 2270302
- [Background] Carter JH, Stewart BJ, Archbold PG, Inoue I, Jaglin J, Lannon M, Rost-Ruffner E, Tennis M, McDermott MP, Amyot D, Barter R, Cornelius L, Demong C, Dobson J, Duff J, Erickson J, Gardiner N, Gauger L, Gray P, Kanigan B, Kiryluk B, Lewis P, Mistura K, Malapira T, Zoog K, et al. Living with a person who has Parkinson's disease: the spouse's perspective by stage of disease. Parkinson's Study Group. Mov Disord. 1998 Jan;13(1):20-8. doi: 10.1002/mds.870130108. PMID 9452321
- [Background] Hudson PL, Hayman-White K. Measuring the psychosocial characteristics of family caregivers of palliative care patients: psychometric properties of nine self-report instruments. J Pain Symptom Manage. 2006 Mar;31(3):215-28. doi: 10.1016/j.jpainsymman.2005.07.010. PMID 16563316
- [Background] Pucciarelli G, Savini S, Byun E, Simeone S, Barbaranelli C, Vela RJ, Alvaro R, Vellone E. Psychometric properties of the Caregiver Preparedness Scale in caregivers of stroke survivors. Heart Lung. 2014 Nov-Dec;43(6):555-60. doi: 10.1016/j.hrtlng.2014.08.004. Epub 2014 Sep 18. PMID 25239706
- [Background] Steffen AM, McKibbin C, Zeiss AM, Gallagher-Thompson D, Bandura A. The revised scale for caregiving self-efficacy: reliability and validity studies. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P74-86. doi: 10.1093/geronb/57.1.p74. PMID 11773226
- [Background] Steffen AM, Gallagher-Thompson D, Arenella KM, Au A, Cheng ST, Crespo M, Cristancho-Lacroix V, Lopez J, Losada-Baltar A, Marquez-Gonzalez M, Nogales-Gonzalez C, Romero-Moreno R. Validating the Revised Scale for Caregiving Self-Efficacy: A Cross-National Review. Gerontologist. 2019 Jul 16;59(4):e325-e342. doi: 10.1093/geront/gny004. PMID 29546334
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Lorig K, Ritter PL, Laurent DD, Yank V. Building Better Caregivers: A Pragmatic 12-Month Trial of a Community-Based Workshop for Caregivers of Cognitively Impaired Adults. J Appl Gerontol. 2019 Sep;38(9):1228-1252. doi: 10.1177/0733464817741682. Epub 2017 Nov 14. PMID 29165000
- [Background] Sarabia-Cobo C, Perez V, de Lorena P, Saenz-Jalon M, Alconero-Camarero AR. Effectiveness of a telephone intervention based on motivational health coaching for improving the mental health of caregivers of people with dementia: A randomised controlled trial. Int J Older People Nurs. 2021 Sep;16(5):e12398. doi: 10.1111/opn.12398. Epub 2021 Aug 1. PMID 34337869
- [Background] Coon DW, Thompson L, Steffen A, Sorocco K, Gallagher-Thompson D. Anger and depression management: psychoeducational skill training interventions for women caregivers of a relative with dementia. Gerontologist. 2003 Oct;43(5):678-89. doi: 10.1093/geront/43.5.678. PMID 14570964
- [Background] 2020 Alzheimer's disease facts and figures. Alzheimers Dement. 2020 Mar 10. doi: 10.1002/alz.12068. Online ahead of print. PMID 32157811
- See also: AARP, National Alliance for Caregiving. Caregiving in the U.S. 2020. AARP; 2020. doi:10.26419/ppi.00103.001 — https://www.aarp.org/pri/topics/ltss/family-caregiving/caregiving-in-the-united-states/
- See also: National Research Summit on Care Services and Supports for Persons with Dementia and Their Caregivers: Report to the National Advisory Council on Alzheimer's Research, Care, and Services.; 2018. — https://aspe.hhs.gov/reports/national-research-summit-care-services-supports-persons-dementia-their-caregivers-final-summit-0
- See also: Reinhard S, Ryan E. Stepping Up to Support Family Caregivers. blog.aarp.org. June 7, 2016. https://blog.aarp.org/thinking-policy/stepping-up-to-support-family-caregivers — https://blog.aarp.org/thinking-policy/stepping-up-to-support-family-caregivers